CLINICAL TRIAL: NCT03156764
Title: The Accuracy of Qp/Qs Calculated by Noninvasive Methods in Children With Shunt Dependent Pulmonary Circulation
Brief Title: Qp/Qs Ratio by Noninvasive Methods in Children With Shunt Dependent Pulmonary Circulation
Status: Terminated | Type: Observational
Why Stopped: More than 100 invasive and non-invasive QpQs data were collected
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: 2017-1046
Record Dates: First submitted 2017-05-10; First posted 2017-05-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia, General; Congenital Heart Disease; Blood Gas Monitoring, Transcutaneous; Blood Gas Analysis
Keywords: Qp/Qs ratio; Pediatric congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Qp/Qs ratio monitoring: Qp/Qs ratio monitoring
  Interventions: Other: Qp/Qs ratio monitoring

INTERVENTIONS:
Other: Qp/Qs ratio monitoring — Op/Qs -monitor will be calculated using SpO2 and cerebral oximetry Op/Qs -blood will be calculated using ABGA and VBGA

SUMMARY:
In pediatric cardiac patients with shunt dependent pulmonary circulation, Qp/Qs ratio is a important parameter indicating the balance of pulmonaty and systemic circulation.

This study will calculate Qp/Qs using variables measured using non-invasive monitors (cerebral oximeter and pulse oximeter). This value will be compared with Qp/Qs calculated using variables obtained from blood sample.

DETAILED DESCRIPTION:
Blood sampling will be performed in both arterial and central venous lines.

ELIGIBILITY:
Inclusion Criteria:

1. pediatric cardiac patients scheduled to cardiac operation (shunt dependent pulmonary circulation)
2. preoperative SpO2<97%

Exclusion Criteria:

1. unable to measure pulse oximeter or cerebral oximeter signal
2. unable to measure SaO2 or SmvO2
3. unstable vital sign

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric cardiac patients scheduled to cardiac operation (shunt dependent pulmonary circulation)
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
the difference between Qp/Qs-monitor and Qp/Qs-blood | within 1 week after surgery
  the difference between Qp/Qs-monitor (measure by pulse oximeter and NIRS) and Qp/Qs-blood (measured by blood gas analysis)

SECONDARY OUTCOMES:
the difference between SpO2 and SaO2 | within 1 week after surgery
  the difference between SpO2 (measure by pulse oximeter)and SaO2 (measured by blood gas analysis)
the difference between cerebral oximeter score and and SmvO2 | within 1 week after surgery
  the difference between cerebral oximeter (measure by NIRS)and SmvO2 (measured by blood gas analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea